CLINICAL TRIAL: NCT03803098
Title: Evaluation of the Metrological Reliability of Connected Objects Available to the Public in the Measurement of Medical Physiological Parameters
Brief Title: Evaluation of the Metrological Reliability of Connected Objects in the Measurement of Medical Physiological Parameters
Acronym: EVALEXPLO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI18035J
Record Dates: First submitted 2018-10-22; First posted 2019-01-14 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Respiratory; Disorder, Functional, Impaired

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: reference measure — measure of a physiological parameter performed with the gold standard medical device
Device: alternative measure — measure of a physiological parameter performed with the connected device under evaluation

SUMMARY:
Many connected objects available over-the-counter to the general public claim to measure physical quantities that may have a medical application. Examples include heart rate, oxygen saturation, respiratory rate, blood pressure, body composition between body fat, lean mass and bone mass, and motion analysis. .

The continuous collection of these quantities by a cheap and easily accessible device opens important medical perspectives in the areas of home monitoring of chronic diseases or preventive medicine in general. Nevertheless, the medical decisions that could be made on the basis of the information provided by these objects require that the measurement be reliable, which is not always the case.

The evaluation of the accuracy of measurements made by these objects therefore seems to be a prerequisite for future use in a medical context. This study therefore proposes to test the adequacy between "gold-standard" measurements carried out in consultation in the department of functional explorations of the Bichat Claude-Bernard hospital and the measurements of the same parameters by connected objects, under the conditions of intended uses by their manufacturer.

DETAILED DESCRIPTION:
Primary objective : Evaluate, in patients consulting for polysomnography, respiratory functional explorations or osteodensitometry, or as part of a day hospital cardiology. The accuracy of the measurement provided by a connected object in relation to the "gold standard" measurement made during the visit. The parameters studied will be:

* For polysomnography, pulse oxygen saturation (SpO2), heart rate (HR) and respiratory rate (RF), sleep quality (efficacy, duration of mild slow sleep, deep slow sleep and REM sleep)
* For bone densitometry, body composition in lean mass, fat mass and bone mass, weight • For respiratory function tests, pulse oxygen saturation (SpO2) and heart rate (HR)
* For day hospitalization in cardiology, blood pressure (BP), heart rate (HR) and heart rate, existence of rhythm disorders or conduction

Secondary objectives:

* Evaluate the ease of use of the device (evaluated by an ad-hoc questionnaire completed by the nursing staff)
* Describe the temporal evolution of the recorded parameters (excluding osteodensitometry for which the measurement is unique)
* For day hospitalization in cardiology, evaluate the diagnostic performance of objects tested on the existence of cardiac rhythm disorders (sinus bradycardia, sinus tachycardia, atrial fibrillation, presence of extrasystoles) or conduction disorders (atrioventricular block). -ventricular, branch block)

ELIGIBILITY:
Inclusion criteria :

* Patient over 18 years old
* Patient sent to the functional exploration department of Bichat hospital to perform one of the following exams: polysomnography, bone densitometry, respiratory function tests, cardiology day hospital assessment
* Patient agreement to participate in the study,
* Affiliated to a social security scheme (benefiting or entitled)

Exclusion criteria :

No defined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred to the physiology department for at least one examination among : polysomnography, bone densitometry, respiratory functino test, day hospital of cardiology.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-02-12 (Estimated); Study Completion 2022-08-12 (Estimated)

PRIMARY OUTCOMES:
relative error between the gold-standard measure of the physiological parameter and the corresponding measure with the tested device, | the two measures are succesive of the day of the examination
  relative error expressed on a percentage

SECONDARY OUTCOMES:
absolute error between the gold-standard measure of the physiological parameter and the corresponding measure with the tested device, | the two measures are succesive of the day of the examination
  absolute error expressed on the unit of the reference measurement

CONTACTS AND LOCATIONS:
Overall Officials: Justine FRIJA MASSON, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Justine Frija, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Frija J, Millet J, Bequignon E, Covali A, Cathelain G, Houenou J, Benzaquen H, Geoffroy PA, Bacry E, Grajoszex M, d'Ortho MP. Proposition of a new, minimally-invasive, software smartphone device to predict sleep apnea and its severity. Sleep Breath. 2025 Sep 5;29(5):282. doi: 10.1007/s11325-025-03441-w. PMID 40911165
- [Derived] Frija-Masson J, Mullaert J, Vidal-Petiot E, Pons-Kerjean N, Flamant M, d'Ortho MP. Accuracy of Smart Scales on Weight and Body Composition: Observational Study. JMIR Mhealth Uhealth. 2021 Apr 30;9(4):e22487. doi: 10.2196/22487. PMID 33929337